CLINICAL TRIAL: NCT06074263
Title: Search to Advance Limited Use of Opioids Pilot: Optimization of Non-Opioid Therapy With a Steroid
Acronym: SAILS-Steroid
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Terminated after 8 participants as prospect for funded is no longer viable
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Cecile A. Feldman, DMD, Dean & Distinguished Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Pro2023001077
Record Dates: First submitted 2023-09-27; First posted 2023-10-10 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Pain Management
Keywords: Pain; Analgesic; Steroid
MeSH Terms: conditions — Agnosia; Pain | interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: Impacted Mandibular 3rd Molar Extraction Model
Who Masked: Participant, Care Provider
Masking Description: Dexamethasone 8mg is being provided in a capsule. The placebo is also being provided in the same capsule.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Steroid (Experimental): Dexamethasone 8mg
  Interventions: Drug: Dexamethasone 8mg
- Placebo (Placebo Comparator): Placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dexamethasone 8mg — Dexamethasone 8mg will be taken orally just prior to surgery.
  Arms: Steroid
Other: Placebo — Placebo capsule which looks identical to dexamethasone capsule
  Arms: Placebo

SUMMARY:
To provide health care professionals, including dentists, with the best possible evidence for clinical decision making when deciding upon analgesics and use of corticosteroid for acute post-surgical pain management; a pilot double blind randomized clinical trial will be conducted to test the hypothesis that use of preemptive dose of corticosteroid will reduce the need for opioid rescue. The impacted 3rd molar extraction model will be used due to the predictable severity of the post-operative pain and generalizability of results, as well as the fact that dentists write about one third of opioid prescriptions for adolescents.

DETAILED DESCRIPTION:
The primary objective of this pilot study is to determine whether a STEROID (1 dose of 8 mg dexamethasone) is superior to CONTROL in pain management and patient satisfaction observed for seven days following 3rd molar extraction, for the relief of acute post-surgical pain.

A double blind, prospective, randomized quasi-pragmatic clinical trial comparing a preemptive dose of 8mg dexamethasone to control will be conducted. Both STEROID and CONTROL will be provided 400 mg ibuprofen and 500 mg acetaminophen as analgesics.

The Research Coordinator will obtain consent with the potential participant followed by a detailed review of inclusion and exclusion criteria. The 3rd molar surgery appointment will occur within 3 months (93) days after obtaining consent, and randomization will occur prior to the 3rd molar extraction procedure. Randomization will be performed within each site, stratified by gender to ensure that randomization procedures will apply equally to men and women. Subgroup analyses will be performed.

The steroid intervention will be administered just prior to surgery, and participants will be followed for 9 (-/+5) days post-surgery during which subjects will take the non-opioid combination analgesics as needed for pain. This represents the time between surgery and the post-operative visit, covering the entire acute pain phase which is normally 7-10 days long. At Visit 1 (Surgery Visit), a pre-surgical saliva sample will be obtained, participants will complete a Pre-Operative Subject Questionnaire addressing pain intensity, pain interference, sleep, and overall satisfaction and a post-surgical saliva sample obtained. During the post-operative period, participants will be asked to complete a diary with morning and evening entries. They will also be asked to collect 8 additional saliva samples: for the first three days just prior to going to sleep and for three day just after getting up in the morning, as well, the night before their post-operative exam and the morning of their post-operative exam. When the participant returns for his/her post-operative visit, generally 7 to 10 days after surgery, he/she will return the pill bottles or blister pack with unused medication and a survey will be administered.

ELIGIBILITY:
Inclusion Criteria:

* Be able to understand the informed consent.

  * Provide signed and dated informed consent form
  * Be able to understand all directions for data gathering instruments in English
  * Be willing and able to comply with all study procedures, including having a smart phone, and be available for the duration of the study
  * Planning to undergo extraction of one or more partial or fully impacted mandibular 3rd molars
  * Be 18 years or older
  * Be in good general health as evidenced by medical history
  * Women must agree to use one of the following methods of contraception while participating in this study:

    * contraceptive pill
    * intra-uterine device
    * condoms
    * abstinence

Exclusion Criteria:

* • History of gastrointestinal bleeding, diverticulitis and/or ulcerative disease

  * History of renal disease (excluding kidney stones)
  * History of hepatic disease
  * History of cardiovascular disease (MI or stroke with the past 6 months)
  * History of bleeding disorder
  * History of Sickle Cell disease
  * Active or untreated asthma
  * History of known allergic reaction to ibuprofen, acetaminophen, or dexamethasone
  * History of myasthenia gravis
  * Currently immunocompromised
  * Currently have a fungal infection
  * Currently taking steroids
  * Currently pregnant or lactating
  * Currently taking CYP3A4 inhibitors

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Pain Experience | 24, 48 and 72 hours
  The arithmetic mean of ratings to four questions -- What is the worst pain, What is the least pain,W is the average pain and How much pain do you feel now on a a numeric rating scale from 0 to 10 where 0 =no pain ) to 10 (the worst pain you can imagine) over the last 12 hours. (Higher number is greater pain)
Satisfaction With Medication | 72 hours
  13 question surveys asking about the participants satisfaction with pain management medication.. Questions ask about pain management, pain interference, and adverse events. Using Likert scales participants are asked how satisfied they are with the (1) ability of the study medication to control their pain, (2) time it took for pain medication to work, (3) amount of pain relief provided by their pain medication, (4) duration of the pain relief provided by their medication, (5) extent side effects interfered with their ability to carry out daily functions, extent side effects affected their cognitive function and (6) extent did side effects affected their mental state. Participants are also asked (1) did their level of pain relief meet their expectations and (2) overall, taking everything into account, how satisfied were they with their study pain medication. The sum of the Likert scale results will be calculated. A higher score indicates greater satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Cecile Feldman, DMD, BMA, Principal Investigator — Rutgers University, School of Dental Medicine
Locations (1):
- Rutgers School of Dental Medicine, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
As this is a pilot study, there is no plan to share data with other researchers.